CLINICAL TRIAL: NCT05031650
Title: Can Open Lung Strategy During Non-Invasive Respiratory Support of Very Premature Infants in the Delivery Room Reduce Non-Invasive Ventilation Failure Compared With Standard Approach? A Randomised Controlled Multicentric Trial
Brief Title: Open Lung Strategy During Non-Invasive Respiratory Support of Very Preterm Infants in the Delivery Room
Acronym: OpenCPAP-DR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Funda Tuzun, Assoc. Prof. Dr., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dokuz Eylul Neonatology
Record Dates: First submitted 2021-08-17; First posted 2021-09-02 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Distress Syndrome in Premature Infant; Non-invasive Ventilation; Lung Injury
Keywords: nasal CPAP; delivery room; open lung strategy; PEEP; Respiratory Distress Syndrome; Individualised ventilation
MeSH Terms: conditions — Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- openCPAP (Active Comparator): Immediately after birth, early nCPAP will be started with a nasal mask with a T-piece resuscitator with 8 cm H2O pressure and 0.30 fiO2. The heart rate (HR) and preductal saturation (SpO2) will be evaluated every 30 seconds. Individually, the following steps will be done according to the situation:
  * If the HR > 120 / min and SpO2 not measured yet or be in the target range: The pressure will be continue as 8 cmH2O.
  * If the HR between 100-120 but SpO2 below the target range or not measured yet : First the pressure will be increased to 10 cm H2O; than fiO2 will be increased gradually if the patient will not respond to 10 cmH2O pressure. Pressure will be reduced to 8 cmH2O if the HR remains> 120 / min and oxygen requirement <0.30 for more than 60 seconds.
  Interventions: Procedure: openCPAP
- standardCPAP (Active Comparator): Immediately after birth, early nCPAP will be started with a nasal mask with T-piece resuscitator at 6 cmH2O pressure and 0.30 fiO2. HR and preductal saturation will be evaluated every 30 seconds. The following steps will be performed according to the situation:
  * If the HR > 120 / min and SpO2 be in the target range or not measurable yet: The pressure will be continue as 6 cmH2O.
  * If the HR between 100-120 but SpO2 below the target range or not measured yet : The pressure will increased up to 8 cm H2O. FiO2 will be increased gradually if the patient will not respond to 8 cmH2O pressure. Pressure will be reduced to 6 cmH2O if the HR remains> 120 / min and oxygen requirement <0.30 for more than 60 seconds.
  Interventions: Procedure: standardCPAP

INTERVENTIONS:
Procedure: openCPAP — Randomized to : Individualized high level CPAP between 8-10 cmH2O pressure
  Arms: openCPAP
Procedure: standardCPAP — Randomized to : Standard level CPAP between 6-8 cmH2O pressure
  Arms: standardCPAP

SUMMARY:
The opening and aeration of the lung is critical for a successful transition from fetal to neonatal life. Early nasal CPAP in the delivery room in spontaneously breathing premature babies with a gestational age of 30 weeks or less is a standard treatment approach since it reduces the need for invasive mechanical ventilation and surfactant therapy. In respiratory distress syndrome (RDS) management, providing optimal lung volumes in the very early period from the beginning of delivery room approaches probably augments the expected lung protective effect. Although the benefits of CPAP support are well known, standart CPAP pressures recommended in the guidelines may not meet the needs of individual babies. Maintaining lung patency in the delivery room is the main mechanism of action of CPAP and the requirement may vary individually depending on lung physiology.

In this multicenter randomized controlled study, we aimed to compare the effects of CPAP therapy applied with a personalized open lung strategy (openCPAP), and standard CPAP therapy (standardCPAP) on oxygenation, respiratory support need and surfactant treatment requirement in preterm babies with RDS in the delivery room.

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 30 completed weeks of gestation and received early nCPAP immediately after birth in delivery room

Exclusion Criteria:

* Requirement of surfactant or endotracheal intubation or positive pressure ventilation before the completion of interventions
* Major congenital anomaly
* Transportation to another hospital

Ages: 1 Minute to 2 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of invasive mechanical ventilation | First 72 hours after the intervention
  Need for intubation and mechanical ventilation (MV) Need for intubation and mechanical ventilation (MV)
Incidence of Surfactant therapy | First 72 hours after the intervention
  Surfactant therapy requirement
SpO2 at 5th minute | 5 minute after the delivery
  The oxygen saturation of the blood at 5 th minute
SpO2 at 10th minute | 5 minute after the delivery
  The oxygen saturation of the blood at 10 th minute

SECONDARY OUTCOMES:
Incidence of pneumothorax | First 24 hours after the intervention
  Incidence of pneumothorax during intervention and within 24 hours
Incidence ofIVH (Grade 3-4) | First 72 hours after the intervention
  Intraventricular hemorrhage (IVH)
Duration of ventilatory support (non-invasive) | During first hospitalisation ( an average of 10 weeks)
  Duration of non-invasive MV (days)
Duration of invasive ventilatory support | During first hospitalisation ( an average of 10 weeks)
  Duration of invasive MV ( days)
Duration of oxygen (O2) | During hospitalisation ( an average of 10 weeks)
  Duration of O2 treatment (days)
Incidence of Surfactant treatment | During hospitalisation (an average of 10 weeks)
  Mean number of surfactant treatment
Bronchopulmonary dysplasia (BPD) | At 36th postnatal week or discharge (an average of 10 weeks after intervention ) whichever came first
  Incidence of BPD
Mortality | through study completion (an average of 10 weeks)
  Death or composite outcome death/BPD

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Ozkan, Prof., Principal Investigator — Dokuz Eylül University- Faculty of Medicine; Nuray Duman, Prof., Study Director — Dokuz Eylül University- Faculty of Medicine; Funda Tuzun, Assoc.Prof., Principal Investigator — Dokuz Eylül University- Faculty of Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik Zubeyde Hanım Maternity and Children Hospital, Ankara
  - Dokuz Eylul University, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duman N, Durukan Tosun M, Tuzun F, Egeli T, Bas AY, Pamukcu MM, Deliloglu B, Akyildiz C, Armagan C, Keskinoglu P, Demirel N, Ozkan H. Non-invasive open lung strategy in delivery room: randomized controlled trial (OpenCPAP-DR). Eur J Pediatr. 2025 Nov 17;184(12):766. doi: 10.1007/s00431-025-06613-8. PMID 41247385